CLINICAL TRIAL: NCT01848951
Title: Comparison of Epidural Analgesia With Bilateral Dual TAP Infiltration Block With Liposomal Bupivacaine in Patients With Major Abdominal Surgery
Brief Title: Comparison of Epidural and TAP Block in Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0287-13-FB
Record Dates: First submitted 2013-04-25; First posted 2013-05-08 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Acute Pain; Surgery; Regional Anesthesia
MeSH Terms: conditions — Acute Pain | interventions — Injections, Epidural; Anesthetics, Local

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Epidural: The skin will be disinfected with 2% chlorhexidine. Under sterile technique, the epidural will be placed. Epidural catheter will be placed at thoracic vertebral levels T5 to T10. Level chosen as clinically indicated. The epidural solution should contain institution's standard solution of Bupivicaine 0.05% and hydromorphone 10 mcg/cc. However, solution type should be clinically indicated.
  Interventions: Drug: Epidural
- TAP Block: The skin will be disinfected with 2% chlorhexidine. The bilateral dual TAP infiltrative blocks will be placed using high-frequency ultrasound. The TAP blocks will be performed using lipospheric bupivacaine (Exparel) with the following dosing regimen.A 266mg (20cc) vial of lipospheric bupivacaine will be equally into 2 30 ml syringes using strict sterile technique. The solution will be diluted in each syringe with 20cc preservative free sterile 0.9% normal saline to a total volume of 30 ml in each syringe. Once the transversus abdominal plane is identified then a 5-10 ml of plain 0.9% normal saline will be injected to open the fascial plane. Once the plane is opened then the 15cc of diluted lipospheric bupivacaine will be administered under direct ultrasound visualization in all 4 TAP quadrants (subcostal position x2 and lateral position x2)
  Interventions: Drug: TAP Block

INTERVENTIONS:
Drug: Epidural — The skin will be disinfected with 2% chlorhexidine. Under sterile technique, the epidural will be placed. Epidural catheter will be placed at thoracic vertebral levels T5 to T10. Level chosen as clinically indicated. The epidural solution should contain institution's standard solution of Bupivicaine 0.05% and hydromorphone 10 mcg/cc. However, solution type should be clinically indicated.
  Other Names: local anesthetic
  Groups: Epidural
Drug: TAP Block — The skin will be disinfected with 2% chlorhexidine. The bilateral dual TAP infiltrative blocks will be placed using high-frequency ultrasound. The TAP blocks will be performed using lipospheric bupivacaine (Exparel) with the following dosing regimen.A 266mg (20cc) vial of lipospheric bupivacaine will be equally into 2 30 ml syringes using strict sterile technique. The solution will be diluted in each syringe with 20cc preservative free sterile 0.9% normal saline to a total volume of 30 ml in each syringe. Once the transversus abdominal plane is identified then a 5-10 ml of plain 0.9% normal saline will be injected to open the fascial plane. Once the plane is opened then the 15cc of diluted lipospheric bupivacaine will be administered under direct ultrasound visualization in all 4 TAP quadrants (subcostal position x2 and lateral position x2)
  Other Names: transversus abdominis plane, abdominal muscle anesthesia
  Groups: TAP Block

SUMMARY:
This study will compare the infiltrative transversusabdominis plane (TAP) block with liposomal bupivacaine to epidural analgesia (EA) in major abdominal surgery . The efficacy of the TAP block for abdominal surgery is well documented in literature, but there are no studies utilizing long-acting bupivacaine. The investigators believe the study will demonstrate no difference between the two in terms of pain scores and opioid consumption, but TAP blocks will decreased costs, urinary retention, and hypotension.

DETAILED DESCRIPTION:
This study intends to examine this rational by comparing the infiltrative transversusabdominis plane (TAP) block with liposomal bupivacaine to EA in major abdominal surgery. The efficacy of the TAP block for abdominal surgery is well documented in the literature, but there are no studies utilizing long-acting bupivacaine. The investigators believe the primary outcome will demonstrate no difference between the two in terms of pain scores and opioid consumption. The investigators anticipate that patients who have undergone TAP blocks will have improved secondary outcomes with respect to a decreased costs, urinary retention, and hypotension.

ELIGIBILITY:
Inclusion Criteria:

* subject >/= 19 years of age
* Undergoing major abdominal surgery
* able to provide written informed consent

Exclusion Criteria:

* chronic opioid use
* allergies to amide anesthetics
* inability to undergo general anesthesia
* pregnancy
* any existence of contraindications to regional anesthesia in the presence of antiplatelet or anticoagulative drugs
* or evidence of gross neurological dysfunction of the lower extremity

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects undergoing major abdominal surgery
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Pain scores | 96 hours post-op
  Comparison of pain scores (0 = no pain to 10 = worst pain possible)
Opioid Consumption in a 24-Hour period | 96 hours post-op
  A comparison of opioid consumption in a 24-Hour period at 96 hours post-op between the interventions

SECONDARY OUTCOMES:
Comparison of 96-hour hospital stay costs | 96 hours post-op
  Comparison of 96-hour hospital stay cost between the interventions
Comparison of urinary failure/catheter acquired infection rates | 96 hours post-op
  Comparison of urinary failure/catheter acquired infection rates between the interventions
Comparison of hypotension rates | 96 hours post-op
  Comparison hypotension rates between the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Nicholas, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States